CLINICAL TRIAL: NCT01614288
Title: A Randomized Clinical Trial to Compare the Effectiveness of High Tibial Osteotomy (HTO) With or Without Arthroscopy of the Knee Joint on Quality of Life, Function, Pain and Swelling for Patients With Medical Compartment Osteoarthritis of the Knee
Brief Title: High Tibial Osteotomy (HTO) With or Without Arthroscopy of the Knee Joint
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Dianne Bryant, Associate Professor, University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FKSMC 2010 - 2
Record Dates: First submitted 2012-06-04; First posted 2012-06-07 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Medial Compartment Osteoarthritis of the Knee
Keywords: HTO; Arthroscopy; Quality-of-Life; Gait Analysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Knee Arthroscopy + HTO (Active Comparator)
  Interventions: Procedure: knee Arthroscopy
- HTO Alone (Active Comparator)
  Interventions: Other: No arthroscopy

INTERVENTIONS:
Procedure: knee Arthroscopy — Patient undergoes a knee arthroscopy and HTO
  Arms: Knee Arthroscopy + HTO
Other: No arthroscopy — Patient undergoes an HTO without knee arthroscopy
  Arms: HTO Alone

SUMMARY:
Participants will be randomized to undergo a High Tibial Osteotomy (HTO) with or without a knee scope. Patients will be tested in the Gait Lab, will fill out quality-of-life questionnaires, and have a clinical evaluation done preoperative and at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* All patients booked for an HTO due to OA
* Grades II to IV severity of OA by radiographic evaluation (Kellgren & Lawrence grade)
* OA of the knee primarily involving the medial compartment

Exclusion Criteria:

* Imaging evidence of significant knee joint pathology that would change the decision to do an HTO
* An arthroscopy of the knee within 2 years of planned surgery
* Active joint or systemic infection,
* Major medical illness that would preclude undergoing surgery,
* Patients who are unwilling or unable to be assessed according to study protocol for two years following surgery
* Major psychiatric illness, developmental handicap or inability to read and understand the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
WOMAC | Preoperatively; 3, 6, 12, 18 and 24 months

SECONDARY OUTCOMES:
The Lower Extremity Functional Scale (LEFS) | Preoperatively; 3, 6, 12, 18 and 24 months
Patient Diary to asses swelling, pain and frequency of analgesic and NSAID use. | Daily x 2 weeks post surgery; Weekly x 3 months
SF-12 | Preoperatively; 3, 6, 12, 18 and 24 months
Gait Testing Procedures | 6, 12 and 24 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Dianne Bryant, PhD, Study Director — The University of Western Ontario
Locations (1):
- London Health Sciences Centre - University Hospital, London, Ontario, Canada